CLINICAL TRIAL: NCT02555319
Title: A Feasibility Study to Evaluate the Safety and Short-term Effectiveness of Implantation of Transcatheter Pulmonary Valve (TPV) for the Treatment of Congenital Heart Disease With Pulmonary Valve Disease
Brief Title: A Feasibility Study to Evaluate the Safety and Short-term Effectiveness of Transcatheter Pulmonary Valve (TPV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPV-001
Record Dates: First submitted 2015-09-09; First posted 2015-09-21 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Defects; Cardiovascular Abnormalities; Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis
Keywords: Pulmonary Valve; Transcatheter Pulmonary Valve; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital; Cardiovascular Abnormalities; Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter Pulmonary Valve (Experimental): Transcatheter Pulmonary Valve (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Transcatheter Pulmonary Valve (TPV)

INTERVENTIONS:
Device: Transcatheter Pulmonary Valve (TPV) — Transcatheter Pulmonary Valve Replacement

SUMMARY:
The purpose of this study is to evaluate the safety and short-term effectiveness of implantation of Transcatheter Pulmonary Valve (TPV) for the treatment of congenital heart disease with pulmonary valve disease.

DETAILED DESCRIPTION:
Diverse congenital heart diseases involving the pulmonary artery, such as Tetralogy of Fallot (TOF) with or without pulmonary atresia, or transposition of the great arteries with pulmonary stenosis, require implantation of an artificial conduit between the right ventricle and the pulmonary artery(PA). Because these conduits finally degenerate and result in pulmonary regurgitation and/or stenosis and progressive right ventricle (RV) dilation and eventual failure, patients need repetitive surgery for conduit revision. Transcatheter pulmonary valve implantation (TPVI) is a less invasive alternative to surgery in patients with dysfunctional right ventricular outflow tract (RVOT). TPV is a large-diameter (up to 28 mm) self-expandable stent with a relatively low profile from a nitinol wire backbone with valve leaflets made from porcine pericardial tissue. The TPV is indicated for use in patients with previous undergone replacement of bioprosthetic valve or conduit due to either pulmonary valve atresia, stenosis, regurgitation or a combination of them and present with dysfunctional RVOT requiring treatment for severe pulmonary regurgitation and/or RVOT conduit obstruction. Consecutive subject data should be collected at discharge, 1, 3, 6 month, and 1-5 years post TPV implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 10 years of age
* Body weight greater than or equal to 30 kilograms
* Pulmonary regurgitation ≥moderate pulmonary regurgitation (PR) (≥3+) or RVOT conduit obstruction with mean gradient >35mmHg by echocardiography
* pulmonary artery annulus or in situ conduit size ≥16 and ≤26mm
* Patient willing to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

* Pre-existing mechanical heart valve in any position
* Obstruction of the central veins (pulmonic bioprosthesis delivery system to the heart)
* Coronary artery compression
* A known hypersensitivity to Aspirin or Heparin
* Immunosuppressive disease
* Active infectious disease (e.g. endocarditis, meningitis)
* Estimated survival less than 6 months
* Female of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Procedural success | 5day
  Procedural success is defined as the TPV implant within desired position, RV-PA peak systolic pressure gradient <35mmHg by catheter, less mild pulmonary regurgitation by angiography, and freedom from explantation of the TPV at 24 hours post-implant.
Hemodynamic functional improvement at 6month | 6 month
  Hemodynamic functional improvement is defined as mean RVOT gradient ≤30 mmHg by continuous wave doppler, and a pulmonary regurgitant fraction <20% by cardiac magnetic resonance (MR).
Procedural / Device related serious adverse events at 6month | 6 month

SECONDARY OUTCOMES:
Hemodynamic function | 5 year
  Hemodynamic function will be measured including peak RVOT pressure gradient, mean RVOT pressure gradient, RV-PA pressure gradient, RV pressure, cardiac output, cardiac index, RV end-diastolic volume by echocardiography, cardiac MR, or catheterization.
Severity of pulmonary regurgitation | 5year
Pulmonary regurgitant fraction | 5year
New York Heart Association (NYHA) functional classification | 5 year
Stent fracture | 5 year
Catheter reintervention on TPV | 5 year
Reoperation | 5 year
Procedural / Device related serious adverse events | 5 year
Death (all cause / procedural / device-related) | 5 year
Other adverse events | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Gi Beom Kim, PhD. MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Haehak-ro Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim GB, Song MK, Bae EJ, Park EA, Lee W, Lim HG, Kim YJ. Successful Feasibility Human Trial of a New Self-Expandable Percutaneous Pulmonary Valve (Pulsta Valve) Implantation Using Knitted Nitinol Wire Backbone and Trileaflet alpha-Gal-Free Porcine Pericardial Valve in the Native Right Ventricular Outflow Tract. Circ Cardiovasc Interv. 2018 Jun;11(6):e006494. doi: 10.1161/CIRCINTERVENTIONS.118.006494. PMID 29871940